CLINICAL TRIAL: NCT04354987
Title: Phase I Clinical Trial to Compare the Pharmacokinetics and Safety of CKD-391 With Co-administration of D090 and D337 in Healthy Adult Volunteers
Brief Title: Compare the Pharmacokinetics and Safety of CKD-391
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 152BE18037
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): R+R+T+T Period 1 : R Period 2 : R Period 3 : T Period 4 : T
  Interventions: Drug: CKD-391 10/10mg; Drug: D090, D337
- Group B (Experimental): R+T+R+T Period 1 : R Period 2 : T Period 3 : R Period 4 : T
  Interventions: Drug: CKD-391 10/10mg; Drug: D090, D337
- Group C (Experimental): T+R+T+R Period 1 : T Period 2 : R Period 3 : T Period 4 : R
  Interventions: Drug: CKD-391 10/10mg; Drug: D090, D337
- Group D (Experimental): T+T+R+R Period 1 : T Period 2 : T Period 3 : R Period 4 : R
  Interventions: Drug: CKD-391 10/10mg; Drug: D090, D337

INTERVENTIONS:
Drug: CKD-391 10/10mg — Drug T: CKD-391 10/10mg(Other Name: Test Drug)
  Other Names: Test Drug (T)
Drug: D090, D337 — D090 and D337 co-administration(Other Name: Reference drug)
  Other Names: Reference Drug (R)

SUMMARY:
phase I clinical trial to compare the pharmacokinetics and safety of CKD-391 with co-administration of D090 and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 45 aged in healthy male adult
2. Subjects in good health as determined by physical exams and medical examinations. No congenital or chronic diseases and no abnormal signs determined by medical examinations.
3. Not abnormal or not clinically significant lab values.
4. Subjects who signed informed consent form with good understandings after explanations by investigators.

Exclusion Criteria:

1. No history or presence of clinically significant diseases.
2. Subjects showing adverse reaction to investigational product
3. Genetic problems in galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption.
4. History of myopathy
5. unable to stop drinking and smoking during clinical trials
6. Subjects who donated whole blood within 60 days or donated component blood within 30 days or received blood transfusion within 30 days
7. History of drug abuse
8. Disagree to contraception
9. Subjects who are in any conditions impossible participating in the clinical trials

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~72hours
  To evaluate pharmacokinetic equivalence of experimental arm comparing Cmax
  1) Atorvastatin, unconjugated ezetimibe(Cmax)
AUCt | 0~72hours
  To evaluate pharmacokinetic equivalence of experimental arm comparing AUCt
  1) Atorvastatin, unconjugated ezetimibe(AUCt)

CONTACTS AND LOCATIONS:
Locations (1):
- Jae-Yong Chung, Gyeonggi-do, Seongnam-si, South Korea